CLINICAL TRIAL: NCT01982773
Title: Effectiveness of a Virtual Hope Box Smartphone App in Enhancing Veterans' Coping With Suicidal Ideation: A Randomized Clinical Trial.
Brief Title: Virtual Hope Box - Effectiveness of a Smartphone App for Coping With Suicidal Ideation
Acronym: VHB-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Telehealth and Technology (U.S. Federal Agency)
Collaborators: The Geneva Foundation (Other); Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 001-W81XWH-10-2-0178; 1334 (Other Grant/Funding Number: Geneva Foundation)
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2017-07

CONDITIONS: Suicidal Ideation; Thoughts of Self Harm; Coping
Keywords: Virtual Hope Box
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual Hope Box Smartphone App (Experimental): Use of the smartphone app, Virtual Hope Box on their personal smartphone
  Interventions: Behavioral: Virtual Hope Box Smartphone App
- EnhancedTreatment As Usual (Active Comparator): Subjects will be issued printed materials guiding them in coping with suicidal thoughts, which include information about coping strategies and emergency contact information.
  Interventions: Behavioral: Enhanced Treatment as Usual

INTERVENTIONS:
Behavioral: Virtual Hope Box Smartphone App — Smartphone app
  Other Names: VHB
  Arms: Virtual Hope Box Smartphone App
Behavioral: Enhanced Treatment as Usual — Printed materials
  Other Names: ETAU
  Arms: EnhancedTreatment As Usual

SUMMARY:
A hope box or self soothing kit is a therapeutic tool employed by clinicians with patients expressing suicidal ideation, significant distress, or otherwise at risk of suicidal or non-suicidal self harm. A "Virtual Hope Box" (VHB) takes the common hope box practice and uses smartphone features to enhance the experience. The rich multimedia features on a smartphone allow more varied options. Furthermore, these devices are already a common repository for user-generated and user-preferred media, which will allow for a highly personalized VHB that is highly portable and always available to a user in distress. We hypothesize that:

1. Patients in the (VHB) intervention condition will demonstrate pre-post reductions in 1) severity of suicidal ideation 2) ability to cope with stressors and 3) increases in perceived reasons for living
2. Patients in the intervention condition will demonstrate greater pre-post reductions in symptoms of suicidal ideation, ability to cope with stressors, and perceived reasons for living compared to patients in the (ETAU) control condition.
3. Patients and clinicians will find VHB to be beneficial and its use readily integrated into practice.

DETAILED DESCRIPTION:
Our overall objective in the proposed study is to assess the impact of a virtual hope-box (VHB) smartphone app on suicidal ideation in veterans undergoing clinical therapy who have recently had suicidal ideation or behavior. We propose to conduct this study in two phases:

Phase 1: Modifying the current VHB-β version of the app to accommodate feedback from pilot study participants. The result will be the VHB V1.0 to be tested in phase 2. This component of the study will be conducted by the T2 group located at Joint Base Lewis-McChord.

Phase 2: Implementing a randomized controlled trial comparing the VHB intervention with enhanced treatment as usual (ETAU) in clinical practice. This component of the study will be conducted at the Portland VA Medical Center.

This research project seeks to answer several essential questions:

1. Can a smartphone app containing the essential components of a hope box and associated elements of CT/DBT (Dialectical Behavioral Therapy) reduce severity of suicidal ideation, and increase perceptions of reasons for living and ability to cope, in a clinical sample of veterans?
2. Is a smartphone VHB app more effective in reducing severity of suicidal ideation, and increasing perceptions of reasons for living and ability to cope, compared to enhanced treatment as usual (ETAU)? In addition, we will gather important information about implementing and integrating VHB as a treatment component in mental health treatment

ELIGIBILITY:
Inclusion Criteria:

* US Service Veterans in active treatment by Portland VA mental health clinicians
* Patients expressing suicidal ideation, thoughts of suicidal self-harm, or determined to be at "high risk" for suicide by treating clinician or Suicide Prevention Team
* Patients owning and regularly using/carrying their own iPhone or Android phones
* Patients identified as clinically suitable by their clinicians for hope box utilization or enhanced treatment as usual (ETAU) as part of treatment

Exclusion Criteria:

* Moderate or severe dementia or significant cognitive disturbance as indicated by chart diagnosis of dementia or score of greater than or equal to 10 on the Short Blessed questionnaire during screening
* Patients considered terminally ill according to documentation in patient records
* Patients with designated guardians, who are unable to provide consent without the assistance of a legally authorized representative or guardian
* Patients admitted to inpatient unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2014-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nigel E Bush, PhD, Principal Investigator — National Center for Telehealth and Technology; Steven K Dobscha, MD, Principal Investigator — Portland VA Medical Center
Locations (2):
- United States (2):
  - Portland VA Medical Center, Portland, Oregon
  - National Center for Telehealth and Technology, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bush NE, Reger MA, Luxton DD, Skopp NA, Kinn J, Smolenski D, Gahm GA. Suicides and suicide attempts in the U.S. Military, 2008-2010. Suicide Life Threat Behav. 2013 Jun;43(3):262-73. doi: 10.1111/sltb.12012. Epub 2013 Jan 17. PMID 23330611
- [Background] Chartrand MM, Frank DA, White LF, Shope TR. Effect of parents' wartime deployment on the behavior of young children in military families. Arch Pediatr Adolesc Med. 2008 Nov;162(11):1009-14. doi: 10.1001/archpedi.162.11.1009. PMID 18981347
- [Background] Luxton DD, Osenbach JE, Regar MA, et al. Department of Defense Suicide Event Report (DoDSER): Calendar Year 2011 Annual Report: National Center for Telehealth and Technology, Defense Centers of Excellence for Psychological Health & TBI (DCOE); 2011
- [Background] Kemp J, Bossarte RM. Suicide Data Report, 2012: Department of Veterans Affairs, Mental Health Services, Suicide Prevention Program; 2012
- [Background] National Violent Death Reporting System. Centers for Disease Control and Prevention http://www.cdc.gov/ViolencePrevention/NVDRS/index.html, 2009
- [Background] Savitsky L, Illingworth M, DuLaney M. Civilian social work: serving the military and veteran populations. Soc Work. 2009 Oct;54(4):327-39. doi: 10.1093/sw/54.4.327. PMID 19780463
- [Background] Congressional testimony of hearing on veteran suicide prevention by panel of experts from the U.S. Department of Veterans Affairs before the U.S. House Veterans' Affairs Subcommittee on Health December 2.2011. U.S. House Veterans' Affairs Subcommittee on Health 2011
- [Background] Borges G, Nock MK, Haro Abad JM, Hwang I, Sampson NA, Alonso J, Andrade LH, Angermeyer MC, Beautrais A, Bromet E, Bruffaerts R, de Girolamo G, Florescu S, Gureje O, Hu C, Karam EG, Kovess-Masfety V, Lee S, Levinson D, Medina-Mora ME, Ormel J, Posada-Villa J, Sagar R, Tomov T, Uda H, Williams DR, Kessler RC. Twelve-month prevalence of and risk factors for suicide attempts in the World Health Organization World Mental Health Surveys. J Clin Psychiatry. 2010 Dec;71(12):1617-28. doi: 10.4088/JCP.08m04967blu. Epub 2010 Aug 24. PMID 20816034
- [Background] Arsenault-Lapierre G, Kim C, Turecki G. Psychiatric diagnoses in 3275 suicides: a meta-analysis. BMC Psychiatry. 2004 Nov 4;4:37. doi: 10.1186/1471-244X-4-37. PMID 15527502
- [Background] Oquendo MA, Galfalvy H, Russo S, Ellis SP, Grunebaum MF, Burke A, Mann JJ. Prospective study of clinical predictors of suicidal acts after a major depressive episode in patients with major depressive disorder or bipolar disorder. Am J Psychiatry. 2004 Aug;161(8):1433-41. doi: 10.1176/appi.ajp.161.8.1433. PMID 15285970
- [Background] Hall RC, Platt DE, Hall RC. Suicide risk assessment: a review of risk factors for suicide in 100 patients who made severe suicide attempts. Evaluation of suicide risk in a time of managed care. Psychosomatics. 1999 Jan-Feb;40(1):18-27. doi: 10.1016/S0033-3182(99)71267-3. PMID 9989117
- [Background] Borges G, Angst J, Nock MK, Ruscio AM, Walters EE, Kessler RC. A risk index for 12-month suicide attempts in the National Comorbidity Survey Replication (NCS-R). Psychol Med. 2006 Dec;36(12):1747-57. doi: 10.1017/S0033291706008786. Epub 2006 Aug 29. PMID 16938149
- [Background] Holma KM, Melartin TK, Haukka J, Holma IA, Sokero TP, Isometsa ET. Incidence and predictors of suicide attempts in DSM-IV major depressive disorder: a five-year prospective study. Am J Psychiatry. 2010 Jul;167(7):801-8. doi: 10.1176/appi.ajp.2010.09050627. Epub 2010 May 17. PMID 20478879
- [Background] Allen JP, Cross G, Swanner J. Suicide in the Army: a review of current information. Mil Med. 2005 Jul;170(7):580-4. doi: 10.7205/milmed.170.7.580. PMID 16130637
- [Background] Blow FC, Bohnert AS, Ilgen MA, Ignacio R, McCarthy JF, Valenstein MM, Knox KL. Suicide mortality among patients treated by the Veterans Health Administration from 2000 to 2007. Am J Public Health. 2012 Mar;102 Suppl 1(Suppl 1):S98-104. doi: 10.2105/AJPH.2011.300441. PMID 22390612
- [Background] Oldham J. PTSD and Suicide. J Psychiatr Pract. 2008 Jul;14(4):195. doi: 10.1097/01.pra.0000327308.50787.45. No abstract available. PMID 18664887
- [Background] Selby EA, Anestis MD, Bender TW, Ribeiro JD, Nock MK, Rudd MD, Bryan CJ, Lim IC, Baker MT, Gutierrez PM, Joiner TE Jr. Overcoming the fear of lethal injury: evaluating suicidal behavior in the military through the lens of the Interpersonal-Psychological Theory of Suicide. Clin Psychol Rev. 2010 Apr;30(3):298-307. doi: 10.1016/j.cpr.2009.12.004. Epub 2009 Dec 13. PMID 20051309
- [Background] Fontana A, Rosenheck R. Traumatic war stressors and psychiatric symptoms among World War II, Korean, and Vietnam War veterans. Psychol Aging. 1994 Mar;9(1):27-33. doi: 10.1037//0882-7974.9.1.27. PMID 8185865
- [Background] Brenner LA, Homaifar BY, Adler LE, Wolfman JH, Kemp J. Suicidality and veterans with a history of traumatic brain injury: precipitants events, protective factors, and prevention strategies. Rehabil Psychol. 2009 Nov;54(4):390-397. doi: 10.1037/a0017802. PMID 19929120
- [Background] Bodner E, Ben-Artzi E, Kaplan Z. Soldiers who kill themselves: the contribution of dispositional and situational factors. Arch Suicide Res. 2006;10(1):29-43. doi: 10.1080/13811110500318299. PMID 16287694
- [Background] Mahon MJ, Tobin JP, Cusack DA, Kelleher C, Malone KM. Suicide among regular-duty military personnel: a retrospective case-control study of occupation-specific risk factors for workplace suicide. Am J Psychiatry. 2005 Sep;162(9):1688-96. doi: 10.1176/appi.ajp.162.9.1688. PMID 16135629
- [Background] Linehan MM. Suicide intervention research: a field in desperate need of development. Suicide Life Threat Behav. 2008 Oct;38(5):483-5. doi: 10.1521/suli.2008.38.5.483. No abstract available. PMID 19014300
- [Background] Rudd MD, Joiner TE, Jobes DA, King CA. The outpatient treatment of suicidality: An integration of science and recognition of its limitations. Professional Psychology: Research and Practice. 1999; 437-446.
- [Background] Beck AT. The current state of cognitive therapy: a 40-year retrospective. Arch Gen Psychiatry. 2005 Sep;62(9):953-9. doi: 10.1001/archpsyc.62.9.953. PMID 16143727
- [Background] Linehan MM, Comtois KA, Brown MZ, Heard HL, Wagner A. Suicide Attempt Self-Injury Interview (SASII): development, reliability, and validity of a scale to assess suicide attempts and intentional self-injury. Psychol Assess. 2006 Sep;18(3):303-12. doi: 10.1037/1040-3590.18.3.303. PMID 16953733
- [Background] O'Neil ME, Peterson K, Low A, et al. Suicide Prevention Interventions and Referral/Follow Up Services: A Systematic Review. Portland, OR: Evidence-based Synthesis Program (ESP) Center Portland VA Medical Center; March 2012 2012.
- [Background] Driscoll KA, Cukrowicz DC, Reardon ML, Joiner TE. Simple treatment for complex problems: A flexible cognitive behavior analysis system approach to psychotherapy Mahwah, New Jersey: Lawrence Erlbaum Associates, Inc.; 2004

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Virtual Hope Box Smartphone App | EnhancedTreatment As Usual
Started | 58 | 60
Completed | 50 | 56
Not Completed | 8 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Hope Box Smartphone App | EnhancedTreatment As Usual | Total
Number analyzed (Participants) | 58 | 60 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 50 | 101
  >=65 years | 7 | 10 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (13.8) | 48.7 (14.3) | 47.6 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 15 | 37
  Male | 36 | 45 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 47 | 50 | 97
  Unknown or Not Reported | 7 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 41 | 44 | 85
  More than one race | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58 | 60 | 118

OUTCOME MEASURES:

1. Primary Outcome: Beck Scale for Suicidal Ideation
Description: measures self-report severity of suicidal ideation during the past week using 21 items. Three factors are assessed: desire for death, preparation for suicide and actual suicide desire. This measure assess an individual's thoughts, attitudes and intentions regarding suicide. Scores could range from 0 - 48. The higher the score indicated the greater risk for suicidal ideation.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Hope Box Smartphone App | EnhancedTreatment As Usual
Number analyzed (Participants) | 58 | 59
units on a scale | 3.31 (2.6) | 3.58 (2.83)

2. Primary Outcome: Beck Scale for Suicidal Ideation
Description: measures self-report severity of suicidal ideation during the past week using 21 items. Three factors are assessed: desire for death, preparation for suicide and actual suicide desire. This measure assess an individual's thoughts, attitudes and intentions regarding suicide. Scores could range from 0 - 48.The higher the score indicated the greater risk for suicidal ideation.
Time Frame: 3 week follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Hope Box Smartphone App | EnhancedTreatment As Usual
Number analyzed (Participants) | 56 | 55
units on a scale | 3.41 (2.64) | 3.33 (2.76)

3. Primary Outcome: Beck Scale for Suicidal Ideation
Description: as for outcome 2
Time Frame: 6 week follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Hope Box Smartphone App | EnhancedTreatment As Usual
Number analyzed (Participants) | 51 | 55
units on a scale | 2.94 (2.59) | 3.02 (2.82)

4. Primary Outcome: Beck Scale for Suicidal Ideation
Description: as for outcome 2
Time Frame: 12 week follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Hope Box Smartphone App | EnhancedTreatment As Usual
Number analyzed (Participants) | 49 | 55
units on a scale | 3.16 (2.7) | 3.2 (2.71)

ADVERSE EVENTS:
Time Frame: From date of randomization until the date of completion, assessed up to 12 weeks
Arm/Group | Virtual Hope Box Smartphone App | EnhancedTreatment As Usual
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/60
Other Adverse Events (participants affected / at risk) | 1/58 | 1/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Virtual Hope Box Smartphone App (N=58) | EnhancedTreatment As Usual (N=60)
enhanced suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
increased depression (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No